CLINICAL TRIAL: NCT02083198
Title: A Comparison of High and Low Chloride Containing IV Fluid Solutions in Patients Undergoing Major Surgery and/or ICU Admission
Brief Title: Effects of IV Chloride Content on Outcomes
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Bax-BSP-HiLoCl
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: SIRS; Balanced Fluids; Plasmalyte
Keywords: hyperchloremic acidosis; balanced fluids; plasmalyte

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High Chloride: Patients receiving .9% sodium choride for resuscitation
- Low chloride: Patients receiving Plasmalyte for resuscitation

SUMMARY:
This observational study evaluates the impact of high and low chloride containing IV fluids on administrative and clinical outcomes. The study uses a large electronic health dataset and examines patients receiving fluid replacement and resuscitation. The hypothesis is that high chloride solutions are associated with adverse outcomes as measured by administrative data and by clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adults meeting SIRS criteria receiving at least 500 mL of fluid replacement on day of SIRS.

Exclusion Criteria:

* Receipt of starches or other colloids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with SIRS needing fluid replacement
Sampling Method: Non-Probability Sample
Enrollment: 1558 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Hospitalization, Expected Length of inpatient stay is approximately 7 days
  Inpatient mortality. Expected Length of inpatient stay is approximately 7 days

SECONDARY OUTCOMES:
Length of Stay | inpatient hospitalization, Expected Length of inpatient stay is approximately 7 days
Acute renal failure | inpatient hospitalization, Expected Length of inpatient stay is approximately 7 days
Infections | inpatient hospitalization, Expected Length of inpatient stay is approximately 7 days
dysrhythmias | inpatient hospitalization, Expected Length of inpatient stay is approximately 7 days
Electrolyte disorders | inpatient hospitalizationExpected Length of inpatient stay is approximately 7 days

OTHER OUTCOMES:
readmission | 30, 60 and 90 day

CONTACTS AND LOCATIONS:
Locations (1):
- Baxter Healthcare, Deerfield, Illinois, United States

REFERENCES:
- [Derived] Shaw AD, Schermer CR, Lobo DN, Munson SH, Khangulov V, Hayashida DK, Kellum JA. Impact of intravenous fluid composition on outcomes in patients with systemic inflammatory response syndrome. Crit Care. 2015 Sep 12;19(1):334. doi: 10.1186/s13054-015-1045-z. PMID 26370823